CLINICAL TRIAL: NCT02367066
Title: A Single Centre, Double-blind, Randomised, Placebo-controlled, Cross-over Phase I Study to Assess the Pharmacodynamics of Oral AR-C165395XX After Administration of Repeated Doses for 3 Days in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Phase I Study to Assess the Pharmacodynamics of Oral AR-C165395XX in Subjects With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: D6420C00001
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: patients; glycaemic control on metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AR-C165395XX + placebo (Experimental): 1st period AR-C165395XX 2nd period placebo
  Interventions: Drug: AR-C165395XX
- Placebo + AR-C165395XX (Placebo Comparator): 1st period Placebo for AR-C165395XX 2nd period AR-C165395XX
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AR-C165395XX — Oral dose of AR-C165395XX (tablets)
  Arms: AR-C165395XX + placebo
Other: Placebo — Oral dose of placebo for AR-C165395XX (tablets)
  Arms: Placebo + AR-C165395XX

SUMMARY:
A study to assess the Pharmacodynamics of oral AR-C165395XX after Administration of Repeated Doses for 3 days in Subjects with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
A Single Centre, Double-blind, Randomised, Placebo-controlled, Cross-over Phase I Study to Assess the Pharmacodynamics of oral AR-C165395XX after Administration of Repeated Doses for 3 days in Subjects with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria

* Provision of informed consent
* Male or female of non-childbearing potential (postmenopausal, and/or have undergone hysterectomy and/or bilateral oophorectomy or salpingectomy/tubal ligation) aged ≥18.
* Patients with HbA1c ≥7.5 but ≤11% at enrolment visit (Visit 1)
* ody mass index >19 to <38 kg/m2
* he fasting plasma glucose should be in the range of 3-14 mmol/L (54-252 mg/dL, nclusive) on the morning of Visit 1.
* Clinical diagnosis of type 2 diabetes mellitus
* Metformin as only anti-diabetic treatment, at least for the last 3 months

Exclusion Criteria:

* History or sign of any clinically significant disease or disorder which, in the opinion f the investigator, may either put the subject at risk because of participation in the sudy, or influence the results or the subject's ability to participate in the study
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) laboratory results >3x upper level of normal range (ULN) Clinical diagnosis of Type 1 diabetes mellitus and/or history of diabetic ketoacidosis or positive Glutamic Acid Decarboxylase Autoantibodies test (GAD antibodies test).
* Patients treated with single Insulin therapy within the last 3 months

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Uribe-Bruce, MD, MCI, Principal Investigator — Profil Institute for Clinical Research, Inc.; Stanko Skrtic, MD, PhD, Study Director — AstraZeneca R&D Mölndal
Locations (1):
- Research Site, Chula Vista, California, United States

REFERENCES:
- [Derived] Skrtic S, Tyrberg B, Broberg M, Ericsson H, Schnecke V, Kjaer M, Hompesch M, Andersson EM, Ryberg E, Aivazidis A, Wennberg Huldt C, Lofgren L, Morrow L, Parkinson J, Ryden-Bergsten T, Watkins E, Sorhede Winzell M. Exploring the insulin secretory properties of the PGD2-GPR44/DP2 axis in vitro and in a randomized phase-1 trial of type 2 diabetes patients. PLoS One. 2018 Dec 17;13(12):e0208998. doi: 10.1371/journal.pone.0208998. eCollection 2018. PMID 30557325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male or female T2DM patients of non-childbearing potential aged >=18 with 7.5<=HbA1c<=11%, 19<BMI<38 kg/m2, fasting plasma glucose in range 3-14 mmol/L and on Metformin as the only anti-diabetic treatment for the last 3 months
Pre-assignment Details: 30 patients were enrolled in the study. 10 of these were screen failures, leaving 20 patients who started the started the study.
Groups:
- AZD1981-Placebo: Sequence AZD1981-Placebo
- Placebo-AZD1981: Sequence Placebo-AZD1981
Period: Overall Study
Arm/Group | AZD1981-Placebo | Placebo-AZD1981
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1981-Placebo | Placebo-AZD1981 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.10 (9.10) | 54.80 (6.80) | 54.00 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 87.28 (18.95) | 87.59 (20.36) | 87.44 (19.14)
Height [Mean (Standard Deviation); unit: cm] | 166.80 (10.70) | 164.90 (12.59) | 165.80 (11.41)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.13 (3.58) | 32.13 (5.37) | 31.63 (4.47)
T2DM disease duration [Mean (Standard Deviation); unit: Years] | 10.30 (4.24) | 8.60 (5.02) | 9.50 (4.61)
Current Metformin Daily Dose [Mean (Standard Deviation); unit: mg] | 1765.00 (473.78) | 1895.00 (390.48) | 1830.00 (427.78)
HbA1c [Mean (Standard Deviation); unit: %] — Percentage of glycosylated hemoglobin, DCCT
  % | 9.50 (1.24) | 9.30 (0.88) | 9.40 (1.06)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint MMTT AUC(0-4h) for Plasma Glucose
Description: MMTT=Mixed Meal Tolerance Test AUC=Area Under Curve
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: One value per subject and treatment. AZD1981 value calculated at Day -1 to Day 3 if subject in sequence AZ1981-Placebo or at Day 6 to Day 9 if subject in sequence Placebo-AZD1981. Placebo value calculated at Day -1 to Day 3 if subject in sequence Placebo-AZD1981 and at Day 6 to Day 9 if subject in sequence AZD1981-Placebo.
Measure: Geometric Mean (Standard Deviation); unit: h*nmol/L
Groups:
- AZD1981: AZD1981, oral tablet
- Placebo: Placebo, oral tablet
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*nmol/L | 0.92 (1.14) | 0.98 (1.09)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 0.94, 80% CI 2-sided [0.90 to 0.98], Standard Error of Mean 0.02

2. Primary Outcome: Change From Baseline to Endpoint MMTT C_max for Plasma Glucose
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: nmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
nmol/L | 0.93 (1.12) | 0.97 (1.09)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 0.96, 80% CI 2-sided [0.92 to 0.99], Standard Error of Mean 0.03

3. Primary Outcome: Change From Baseline to Endpoint GGI AUC(1-2h) for Plasma C-Peptide
Description: GGI=Glucose and GLP1 infusion AUC=Area Under Curve
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*pmol/L | 1.05 (1.17) | 1.06 (1.20)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.41, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 0.99, 80% CI 2-sided [0.96 to 1.03], Standard Error of Mean 0.03

4. Secondary Outcome: Change From Baseline to Endpoint MMTT AUC(0-4h) for Plasma Insulin
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*mU/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*mU/L | 0.99 (1.23) | 1.08 (1.16)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 0.92, 80% CI 2-sided [0.85 to 0.99], Standard Error of Mean 0.05

5. Secondary Outcome: Change From Baseline MMTT AUC(0-4h) for Plasma Glucagon
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*pmol/L | 1.02 (1.19) | 0.96 (1.25)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 1.06, 80% CI 2-sided [0.99 to 1.13], Standard Error of Mean 0.04

6. Secondary Outcome: Change From Baseline to Endpoint MMTT AUC(0-4h) for Plasma C-Peptide
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*pmol/L | 1.01 (1.15) | 1.09 (1.14)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 0.93, 80% CI 2-sided [0.89 to 0.98], Standard Error of Mean 0.04

7. Secondary Outcome: Change From Baseline to Endpoint GGI AUC(0-1h) for Plasma Insulin
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*mU/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*mU/L | 1.01 (1.19) | 1.07 (1.35)

8. Secondary Outcome: Change From Baseline to Endpoint GGI AUC(1-2h) for Plasma Insulin
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*mU/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*mU/L | 1.03 (1.25) | 1.04 (1.27)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis — 1-sided; Geometric LS MEan Ratio = 1.00, 80% CI 2-sided [0.91 to 1.06], Standard Error of Mean 0.05

9. Secondary Outcome: Change From Baseline to Endpoint GGI AUC(0-1h) for Plasma Glucagon
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*mmol/L | 1.01 (1.08) | 0.97 (1.06)

10. Secondary Outcome: Change From Baseline to Endpoint GGI AUC(1-2h) for Plasma Glucagon
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*mmol/L | 1.01 (1.06) | 0.99 (1.06)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis — 1-sided; Geometric LS Mean Ratio = 1.02, 80% CI 2-sided [1.00 to 1.04], Standard Error of Mean 0.01

11. Secondary Outcome: Change From Baseline to Endpoint Fasting Beta-cell Responsiveness
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 10^-9*(L/kg)*min
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
10^-9*(L/kg)*min | 0.01 (0.01) | -0.00 (0.01)
Statistical Analysis 1: Comparison: AZD1981 vs Placebo; Test type: Superiority or Other; p = 0.45, Mixed Models Analysis — 2-sided; LS Mean Difference = 0.01, 90% CI 2-sided [-0.01 to 0.03], Standard Error of Mean 0.01

12. Secondary Outcome: Fasting Insulin at Endpoint
Time Frame: Day 3 and Day 9
Population: One value per subject and treatment. AZD1981 value calculated at Day 3 if subject in sequence AZD1981-Placebo or at Day 9 if subject in sequence Placebo-AZD1981. Placebo value calculated at Day 3 if subject in sequence Placebo-AZD1981 or at Day 9 if subject in sequence AZD1981-Placebo.
Measure: Least Squares Mean (Standard Error); unit: UIU/ML
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
UIU/ML | 11.70 (1.48) | 11.40 (1.48)

13. Secondary Outcome: Maximum Plasma AZD1981 Concentration at Steady-State, C_ss,Max
Time Frame: Days 2,3,8,9
Population: One value per subject and method (MMTT/GGI). Value calculated on days 2 and 3 if subject in sequence AZD1981-Placebo or on days 8 and 9 if subject in sequence Placebo-AZD1981.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- MMTT: MMTT (Mixed Meal Tolerance Test)
- GGI (Graded Glucose and GLP1 Infusion): GGI (Graded glucose and GLP1 infusion)
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
nmol/L | 2507 (71.09) | 3662 (86.90)

14. Secondary Outcome: Time of Maximum Plasma AZD1081 Concentration, t_ss,Max
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Median (Full Range); unit: h
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 2.00]

15. Secondary Outcome: Plasma AZD1981 AUC(0-1h)
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h*nmol/L | 701.30 (122.30) | 2061 (74.66)

16. Secondary Outcome: Plasma AZD1981 AUC(0-2h)
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Groups:
- MMTT: Mixed Meal Tolerance Test (MMTT)
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h*nmol/L | 2071 (97.56) | 5016 (75.91)

17. Secondary Outcome: Minimum Plasma AZD1981 Concentration at Steady-State, C_ss,Min
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
nmol/L | 202.40 (39.12) | 376.20 (83.28)

18. Secondary Outcome: Plasma AZD1981 AUC(1-2h)
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h*nmol/L | 1344 (88.76) | 2936 (78.72)

19. Secondary Outcome: Plasma Paracetamol Maximum Concentration, C_max
Time Frame: Days 3,9
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
ng/mL | 8074 (37.32) | 7899 (30.51)

20. Secondary Outcome: Time of Maximum Plasma Paracetamol Concentration, t_max
Time Frame: Days 3,9
Population: as for outcome 12
Measure: Median (Full Range); unit: h
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h | 3.50 [0.50 to 4.00] | 3.50 [1.00 to 4.02]

21. Secondary Outcome: Plasma Paracetamol AUC(0-t)
Time Frame: Days 3,9
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/ML
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*ng/ML | 19730 (46.64) | 18850 (26.38)

22. Secondary Outcome: Change From Baseline to Endpoint GGI AUC(0-1h) for Plasma C-Peptide
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*pmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*pmol/L | 1.02 (1.16) | 1.03 (1.18)

23. Secondary Outcome: Change From Baseline to Endpoint GGI AUC(0-24h) for Plasma Glucose
Time Frame: Day -1 to Day 3 and Day 6 to Day 9
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: h*mmol/L
Arm/Group | AZD1981 | Placebo
Number analyzed (Participants) | 20 | 20
h*mmol/L | 0.96 (1.09) | 0.97 (1.08)

24. Secondary Outcome: Plasma AZD1981 AUC(0-4h)
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h*nmol/L | 5793 (53.96) | NA (NA) — PK not measured for this time interval

25. Secondary Outcome: Plasma AZD1981 AUC(0-12h)
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h*nmol/L | 12460 (36.79) | NA (NA) — PK not measured for this time interval

26. Secondary Outcome: Plasma AZD1981 AUC(0-24h)
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
h*nmol/L | 24930 (36.79) | NA (NA) — PK not measured for this time interval

27. Secondary Outcome: Apparent Oral Plasma AZD1981 at Steady-State, CL_ss/F
Time Frame: Days 2,3,8,9
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MMTT | GGI (Graded Glucose and GLP1 Infusion)
Number analyzed (Participants) | 20 | 20
L/h | 21.94 (8.19) | NA (NA) — PK not measured for this time interval

ADVERSE EVENTS:
Arm/Group | AZD1981 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 5/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 (N=20) | Placebo (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 2 | 2
Local swelling (General disorders) | 0 | 1
Vessel puncture site reaction (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No